CLINICAL TRIAL: NCT03413644
Title: Evaluation of ClearLLab Leukemia and Lymphoma Panels
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B88558
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Leukemia-Lymphoma
Keywords: Hematological diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: Flow Cytometry — Immunophenotyping of residual clinical samples tested with ClearLLab diagnostic reagent on a specified Flow Cytometer

SUMMARY:
Multi-center study of specimens from subjects presenting to the flow cytometry laboratory as part of their standard of care for hematological diseases work-up.

DETAILED DESCRIPTION:
Multi-center study of specimens from subjects presenting for flow cytometry immunophenotyping as part of their standard of care for hematological diseases work-up. Residual specimens will be tested using the ClearLLab Panels to determine the presence or absence of an abnormal phenotype and compare results to clinical impression (hematological malignancy or non-malignancy).

ELIGIBILITY:
Inclusion Criteria:

* Residual samples from patients with hematological abnormalities being evaluated by Flow Cytometry for the presence or absence of an abnormal population associated with a hematological malignancy. All subjects of any ethnicity, age and racial background will be included.

Exclusion Criteria:

* Specimens and/or spent samples that are visibly hemolyzed
* Specimens and/or spent samples that are visibly clotted
* Specimens and/or spent samples collected in K2EDTA anticoagulant older than 24 hours from time of collection
* Specimens and/or spent samples collected in Heparin or ACD anticoagulant older than 48 hours from time of collection
* Samples with insufficient volume to complete the protocol tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specimens from new cases or follow up patients suspected of having a hematological malignancy and present with symptoms based on Bethesda guidelines.
Sampling Method: Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Hematologically Malignant or Non-Malignant | Residual samples must be tested within 24 hours of collection in K2EDTA or within 48 hours of collection in Heparin or ACD anticoagulants
  Presence or absence of an abnormal phenotype detected using the ClearLLab Panels vs. the clinical outcome of "Hematologically Malignant" or "Hematologically Non-Malignant" from the same subject

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Padurean, MD, Principal Investigator — NeoGenomics Laboratories, Inc.; Mike Keeney, Principal Investigator — London Health Sciences Center; Joanne Luider, Principal Investigator — Calgary Laboratory Services; Wolfgang Kern, Principal Investigator — Munich Leukemia Laboratory
Locations (4):
- NeoGenomics Laboratories, Inc., Fort Myers, Florida, United States
- Canada (2):
  - Calgary Laboratory Services, Calgary, Alberta
  - London Health Sciences Center, London, Ontario
- Munich Leukemia Laboratory, Munich, Germany